CLINICAL TRIAL: NCT06385249
Title: An Uncontrolled, Prospective, Multicenter, Post-market Clinical Investigation to Confirm the Performance and Safety of Navina Mini, a New CE-marked Low-volume Trans-anal Irrigation (TAI) Device in Children and Adolescents
Brief Title: An Evaluation of Navina Mini, a New Trans-anal Irrigation (TAI) Device in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAV-0012
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Experimental): The subjects are children and adolescents with anal incontinence or bowel outlet problems and deemed suitable for and in need of low-volume TAI as assessed by the investigator.
  Interventions: Device: Navina Mini

INTERVENTIONS:
Device: Navina Mini — Trans-anal irrigation (TAI) with a new CE-marked device, Navina Mini
  Other Names: Trans-anal irrigation (TAI)

SUMMARY:
The study is designed to deliver further information on clinical benefit, patients' satisfaction, and perception of handling and to confirm safety of Navina Mini when used in children and adolescents.

DETAILED DESCRIPTION:
This is an uncontrolled, prospective, multicentre post-market clinical follow-up investigation that will enroll male and female children /adolescents with a need for low-volume transanal irrigation (TAI) as judged by the investigator or designee.

A total of 27 subjects in need of low-volume TAI will be recruited from 2-3 sites in Sweden and will be treated with Navina Mini as per product intended purpose and per instruction of use. Participating subjects will perform three visits during the clinical investigation and will be followed for a total of four (4) to six (6) weeks.

The study is designed to deliver further information on clinical benefit, patients' satisfaction, and perception of handling and to confirm device safety when used in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male and female children/adolescents between 3 and 17 years of age at the time of inclusion
* Diagnosis of at least one of the following:

  * functional constipation not well treated with oral laxatives
  * functional fecal incontinence, either retentive or non-retentive (FNRFI: Functional Non-Retentive Fecal Incontinence) not well treated with oral laxatives
  * neurogenic bowel dysfunction due to spinal abnormalities and/or spinal cord injury or cerebral palsy
  * patient with sequelae of anorectal malformations to Hirschsprung disease
  * Fecal Incontinence (FI) due to iatrogenic injury including tumor surgery sequelae
* Symptom duration of > 3 months
* Subject and/or their legally designated representative can communicate in written and oral Swedish language

Exclusion Criteria:

* Children/adolescents previously treated with, or currently in need of, high volume TAI, i.e., volume > 250 ml
* Confirmed pregnancy at the time of enrollment
* Participating in another clinical investigation interfering with this investigation
* Subjects with an active, symptomatic, inflammatory bowel disease, radiation proctitis, and or active perianal fistula disease
* Rectal bleeding of uncertain origin or active hemorrhoidal bleeding
* < 6 months after anal or colorectal surgery
* Ongoing anti-coagulant therapy (i.e., NOACS, heparin, warfarin)
* Ischemic colitis
* Active anal fissure
* Inability to use the product or anyone to assist in its usage (hand function assessment)
* Person not suitable for the investigation according to the investigator's judgment

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction | up to 6 weeks
  Overall patient satisfaction measured with a 5-graded assessment scale (Patient Reported Outcome (PRO) via Wellspect Questionnaire: 0 = Not at all satisfied, 1 = Not satisfied, 2 = Neither satisfied nor unsatisfied, 3=Satisfied, 4 = Very satisfied)

SECONDARY OUTCOMES:
Incomplete bowel emptying | up to 6 weeks
  Subjects' perception of incomplete bowel emptying measured with a 4-graded assessment scale (PRO via Wellspect Questionnaire: 0 = Never, 1= Seldom, 2= Often, 3= Always)
Episodes of fecal incontinence | up to 6 weeks
  Episodes of obstructed defecation outlet syndrome or episodes of fecal incontinence as documented in a diary on a daily basis
Level of independence | up to 6 weeks
  Patients population able to use the device themselves: need support during the whole procedure, need support in parts of the procedure, no support needed: Yes and No answers
Perception of handling of the device | up to 6 weeks
  Subjects' perception of handling of the device measured with a 5-graded assessment scale (PRO via Wellspect Questionnaire: Evaluation of Navina Mini (0 = Very difficult, 1 = Difficult, 2 = Neither difficult nor easy, 3= Easy, 4 = Very easy) or (0 = Strongly disagree, 1 = Agree, 2 = Neither agree nor disagree, 3 = Agree, 4 = Strongly agree))
Safety outcome | up to 6 weeks
  Assessment of adverse events and device deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wide, Principal Investigator — H.K.H. Kronprinsessan Victorias Barn- och ungdomssjukhus Universitetssjukhuset
Locations (1):
- H.K.H. Kronprinsessan Victorias Barn- och ungdomssjukhus Universitetssjukhuset, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No